CLINICAL TRIAL: NCT03071510
Title: IO-CTNG: A Multi-Centre Evaluation of the Atlas Genetics io® CTNG System Used in Centralised and Point of Care Settings
Brief Title: Evaluation of the Atlas Genetics io® CTNG System
Acronym: IO-CTNG
Status: Completed | Type: Observational
Sponsor: Binx Health Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: MOB-VTP-001
Record Dates: First submitted 2017-02-27; First posted 2017-03-07 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Chlamydia Trachomatis; Gonorrhea
MeSH Terms: conditions — Gonorrhea

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Atlas Genetics io® system — Specimen Collection

SUMMARY:
Atlas Genetics io® system results are compared with those obtained from comparator devices.

DETAILED DESCRIPTION:
Results from the Atlas Genetics io® system are compared with a Composite Infection Status obtained from testing on three commonly used comparator devices.

This is a prospective, single-arm, multi-centre investigation enrolling up to 12,000 adult participants over 14 years of age who are undergoing testing for the presence of CT/NG.

ELIGIBILITY:
Inclusion Criteria:

1. Symptomatic and asymptomatic individuals ≥14 years of age

Exclusion Criteria:

1. Treatment with antibiotics known to be effective against Chlamydia trachomatis and/or Neisseria gonorrhoeae within the previous 4 weeks before inclusion in the study.
2. Unable to self-obtain a vaginal swab or urine sample of at least 30 mL

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Participants over 14 years of age for whom testing for Chlamydia trachomatis and/or Neisseria gonorrhoeae is appropriate
Sampling Method: Probability Sample
Enrollment: 7128 (Actual)
Dates: Start 2017-05-18 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-08-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy compared to positive Composite Infected Status from comparator devices | Up to 7 days
  The assessment of the diagnostic accuracy of the study device as compared to positive Composite Infected Status from comparator devices

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Van der Pol, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (10):
- United States (10):
  - University of Alabama, Birmingham, Alabama
  - AIDS Healthcare Foundation, Los Angeles, California
  - Indiana University, Indianapolis, Indiana
  - Louisiana State University, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - University of Mississippi, Jackson, Mississippi
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest Center for Reproductive Medicine, Greensboro, North Carolina
  - Planned Parenthood Southeastern Pennsylvania, Philadelphia, Pennsylvania
  - Planned Parenthood Gulf Coast, Houston, Texas

IPD SHARING:
Plan to Share IPD: No